CLINICAL TRIAL: NCT07304622
Title: Comprehensive Assessment of the Impact of Various Therapeutic Methods on Gait Quality, Physical and Mental Fitness of Postmenopausal Women.
Brief Title: Impact of Various Therapeutic Methods on Gait Quality, Physical and Mental Fitness of Postmenopausal Women.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The President Stanisław Wojciechowski State University of Applied Sciences in Kalisz (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: Kalisz 2025-09
Record Dates: First submitted 2025-12-01; First posted 2025-12-26 (Actual); Last update posted 2025-12-26 (Actual); Status verified 2025-12

CONDITIONS: Physical Performance and Fitness in Old Age
Keywords: activity in geriatrics; postmenopausal mental fitness; body stability in old age; postmenopausal physical fitness; fullerton test; spirometry

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Coordination Group, the goal is to improve motor coordination and balance (Active Comparator): Eye-hand coordination exercises, balance exercises, walking and running exercises, exercises with scarves and balls, senomotor exercises
  Interventions: Other: Coordination Training
- Mobility Group, the goal is to improve the range of motion in the joints (Active Comparator): Exercisec focused on the mobility of a single joint. The exercises performed in various positions and using small sports equipment. Yoga elements and breathing exercises were also included.
  Interventions: Other: Mobility Training
- Core Stability Group, the goal is to improve postural stability (Active Comparator): Exercises focused on the postural stabilization, exercises for steady positioning while sitting, standing, or moving. The exercises in various positions and using small sports equipment for the balance and core strength
  Interventions: Other: Core Training
- Control Group not participating in any sports activity (No Intervention): The group included 25 women over 65 years of age. The group participated in no sports activities

INTERVENTIONS:
Other: Coordination Training — The group included 25 women over 65 years of age. The group participated in sports activities twice a week for three months. Each training session lasted 45 minutes and focused on the coordination and balance. The exercises were performed in various positions and using small sports equipment to achieve smooth, accurate, and controlled movements.
  These was achieved by exercises with:
  * Coordination ladders - developing rhythm, speed, and precision
  * Unstable surface exercises - improving balance and postural control
  * Reaction exercises (e.g., responding to auditory/visual signals).
  * Multitasking tasks - combining physical and mental elements
  * Exercises in variable conditions (e.g., closed eyes, non-standard equipment).
  * Movement games and activities - varying directions, speeds, and reactions to external stimuli, developing the ability to switch and adapt movement.
  Arms: Coordination Group, the goal is to improve motor coordination and balance
Other: Core Training — The group included 25 women over 65 years of age. The group participated in sports activities twice a week for three months. Each training session lasted 45 minutes and focused on the postural stabilization to keep the body's center of mass within its, allowing for steady positioning while sitting, standing, or moving. The exercises were performed in various positions and using small sports equipment. exercises were chosen to improve the body's ability to control and maintain its position against gravity, enhancing balance and core strength
  Arms: Core Stability Group, the goal is to improve postural stability
Other: Mobility Training — The group included 25 women over 65 years of age. The group participated in sports activities twice a week for three months. Each training session lasted 45 minutes and focused on the mobility of a single joint. The exercises were performed in various positions and using small sports equipment. Yoga elements and breathing exercises were also included.
  Arms: Mobility Group, the goal is to improve the range of motion in the joints

SUMMARY:
The goal of this clinical trial is to learn which physical activity affects the quality of gait, physical and mental fitness of older women. The main questions it aims to answer are:

Does any of the training methods improve the physical or mental fitness of postmenopausal women? Which of these training methods improves the physical and mental condition of postmenopausal women the most?

Researchers will compare the results of three training groups to each other and to control group (with no training) to see which training method has the greatest impact on improving the quality of gait, physical fitness and mental health of postmenopausal women.

Participants took part in physical activity classes that took place for 12 weeks, twice a week for 45 minutes.

Before starting the first and after completing the last physical activity, participants participated in the following tests: resting circulatory parameters, anthropometric tests, respiratory spirometry, cardiorespiratory fitness assessment, Fullerton test, measurement of force distribution and foot pressure, physical activity level assessment (IPAQ), and questionnaires on health-related quality of life (SF-36), geriatric depression scale (GDS), and cognitive function assessment scale (MoCA).

DETAILED DESCRIPTION:
The study aims to comprehensively evaluate three therapeutic methods and their impact on gait quality, physical fitness, and mental well-being. It will allow for the identification of gait patterns, the determination of parameter values separately for the left and right legs, enabling the assessment of gait symmetry, and may indicate injury or pain in the subject, even if these are not yet visible to the observer.

The study group consisted of 100 women over 65 years of age. Each of the three therapeutic methods was represented by 25 participants. The control group, which received no intervention, also consisted of 25 participants. Participants eligible for the project must have no health contraindications to participating in physical activity. Participation in the project is voluntary, and participants may withdraw from participation at any stage.

The three therapeutic methods (interventions) are:

* "Mobility" (with yoga elements) - aimed at improving joint range of motion
* "Coordination and Balance" - aimed at improving motor coordination and balance
* "Core Stability" - aimed at strengthening abdominal, back, and hip muscles

Before the first and after the last exercise class, the following tests was performed:

* resting circulatory system measurements (blood pressure and heart rate),
* anthropometric tests Basic anthropometric measurements was taken (height, weight, selected circumferences, and measurements of the length and width of the trunk and limbs, and a body mass index (BMI) was calculated). Body composition was analyzed. Water content was measured using the bioimpedance method (BIA), which involves passing a very low-intensity, high-frequency current through the human body. The test was performed using a TANITA MC-980 MA device (TANITA, Japan). The test provides information on total body water (TBW), extracellular water (ECW), and intracellular water (ICW). The test is completely non-invasive.
* respiratory spirometry It was performed using the Italian-made MicroQuark device by COSMED; for this purpose, in a sitting position, the women performed three tests during which static and dynamic spirometric parameters will be measured, such as: vital capacity (VC), expiratory reserve volume (ERV), tidal volume (VT), forced vital capacity (FVC), forced expiratory volume in the first second (FEV1), and the Tiffeneau index (FEV1/FVC); minute ventilation (VE) and maximum voluntary minute ventilation (MVV) will also be measured.
* Fullerton test

It was used for a multidimensional assessment of physical fitness. It allows for the observation of gradual decline in fitness with age and assesses tolerance, strength, and flexibility of the upper and lower body, as well as agility and balance. The Fullerton Test consists of six sequentially performed parts:

Arm Curl Test Back Scratch Test 30-Second Chair Stand Chair Sit-and-Reach Test 8-Foot Up-and-Go Test 6-Minute Walk Test

* measurement of force distribution and foot pressur (Lateral balance, foot force and load) Measurements of foot force and pressure distribution was made using a Tekscan MatScan measuring mat with built-in sensors. The test was performed dynamically to identify gait asymmetries. Participants walked across the mat three times with each bare foot to identify differences in the load profiles of the right and left feet, as well as to analyze the dynamics of body weight shift and local high-pressure points. Foot function was also be analyzed by stance phase region. The test is completely non-invasive.
* The International Physical Activity Questionnaire (IPAQ), long version (IPAQ) - Polish version 53 was used to assess physical activity levels. Questions concern physical activity over the last 7 days, including activities performed at work, at home and around the home, while traveling, and during free time devoted to recreation, exercise, or sports.
* questionnaires on health-related quality of life (SF-36) Health-related quality of life was assessed using the SF-36 questionnaire. This questionnaire consists of 36 questions that fall into eight categories related to mental and physical health: physical functioning, health problems limiting the performance of current social functions (physical role), somatic pain, general health, vitality, social functioning, emotional problems limiting the performance of current social functions (emotional role), and mental health.
* geriatric depression scale (GDS) It consists of 30 questions, each answered with a yes or no. If the participant has difficulty understanding the questions, assistance with reading and completing the scale is acceptable. The scale score does not constitute a diagnosis of depression, but it can provide diagnostic guidance.
* The Montreal Cognitive Assessment (MoCA) It is screening tool for detecting mild cognitive impairment (MCI) and early signs of dementia. It assesses multiple cognitive domains, including memory, language, attention, visuospatial skills, executive functions, and orientation, by requiring individuals to perform a series of tasks like drawing a clock face, recalling words, and solving simple math problems.

The study will determine gait patterns and any asymmetries. This information can be useful in selecting potential orthopedic equipment and appropriate corrective exercises.

The prevention of injuries related to falls caused by abnormal gait patterns will be discussed.

The study results will be used to implement therapeutic programs aimed at correcting identified functional abnormalities in older adults. After completing the project, the women participating in the study will receive an exercise program to correct their individual deficits.

ELIGIBILITY:
Inclusion Criteria:

* female
* minimum age 65 years
* independence in performing everyday activities
* ability to actively participate in sports activities twice a week
* consent from the doctor to participate in sports activities

Exclusion Criteria:

* diseases of the locomotor system preventing independement movement
* active or post cancerous disease
* unstable ischemic heart disease
* drug and alcohol addiction

Min Age: 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 100 (Actual)
Dates: Start 2024-10-01 (Actual); Primary Completion 2025-04-11 (Actual); Study Completion 2025-04-30 (Actual)

PRIMARY OUTCOMES:
Level of Physical Fitness | From enrollment to the end of treatment/training at 14 weeks
  physical fitness measured using the Fullerton test
Quality of Life Assessment | From enrollment to the end of treatment/training at 14 weeks
  SF-36 Questionnaire
  * The recoded values for items within a domain are summed and then transformed to a 0-100 scale (0 = worst, 100 = best health).
  * Eight Scales (Domains):
  Physical Functioning (PF) Role Limitations due to Physical Health (RP) Role Limitations due to Emotional Problems (RE) Vitality (VT) Emotional Well-being (MH) Social Functioning (SF) Bodily Pain (BP) General Health (GH)
Assessment of Lung Function | From enrollment to the end of treatment/traing at 14 weeks
  Vital Capacity in liters (L)
Assessment of Lung Function | From enrollment to the end of treatment/traing at 14 weeks
  Tidal Volume in millliliters (mL)
Assessment of Lung Function | From enrollment to the end of treatment/traing at 14 weeks
  Respiratory Rate (RR) in breath per minute (bpm)
Assessment of Lung Function | From enrollment to the end of treatment/traing at 14 weeks
  Tiffeneau-Pinelli Index - FEV1/FVC Ratio (%)
Assessment of Lung Function | From enrollment to the end of treatment/traing at 14 weeks
  Maximal Mid-Expiratory Flow Rate (MMEF or FEF 25-75) in L/s
Level of Physical Fitness | From enrollment to the end of tratment/training at 14 weeks
  IPAQ international physical activity questionnaire (MET-minutes/week units) Measured various domains of the eve-ry-day life: at work, while traveling, doing housework or leisure activities and sports. It mea-sures the time spent sitting at weekdays and weekends. It allows easy classification of the respondents physical activity into three categories: low (below 600 MET-minutes/ week), moderate (600-1500 lub 600-3000 MET-minutes/week) and high (above 1500 or 3000 MET-minutes/week).
Quality of Life Assesment | From enrollment to the end of treatment/training at 14 weeks
  The Geriatric Depression Scale (GDS)
  * scoring involves answering yes/no questions, with points given for specific answers
  * For the common 30-item scale, scores usually mean: 0-9 Normal, 10-19 Mild Depression, 20-30 Severe Depression

SECONDARY OUTCOMES:
Anthropometric Measurements using TANITA MC-980 MA device (TANITA, Japan). | From enrollment to the end of treatment/training at 14 weeks
  The examination was be performed using a TANITA MC-980 MA device (TANITA, Japan), using Bioelectrical Impedance Analysis (BIA)
  - total body water (TBW), extracellular water (ECW), intracellular water (ICW)
Assessment of Cognitive Function | From enrollment to the end of treatment/training at 14 weeks
  Montreal Cognitive Assessment (MoCa) assesses:
  Memory, Attention and concentration, Language, Visuospatial skills, Executive functions, Conceptual thinking and Orientation
  - scoring up to 30 points, with higher scores indicating better function (normal is ~26+)
FootMat Clinical 7.10 Measurement of Foot Load and its Behavior while Walking by pressure sensor mat, MobileMat, provide by Tekscan | From enrollment to the end of treatment/training at 14 weeks
  Metatarsal or Heel Maximum Force in Newton (N)
  1st and 2nd Peak of Foot (left and right) in seconds Measurement of the maximum force and average pressure on the plantar side of the foot while walking (dynamic test)
Antropometric Measurements using TANITA MC-980 MA device (TANITA, Japan) | from enrollment to the end of treatment/training at 14 weeks
  The examination was be performed using a TANITA MC-980 MA device (TANITA, Japan), using Bioelectrical Impedance Analysis (BIA)
  - weight in kiligrams
Anthropometric Measurements using TANITA MC-980 MA device (Tanita, Japan) | from enrollment to the end of treatment/training at 14 weeks
  The examination was be performed using a TANITA MC-980 MA device (TANITA, Japan), using Bioelectrical Impedance Analysis (BIA)
  - BMI - weight and height will be combined to report BMI in kg/m^2
Anthropometric Measurements using TANITA MC-980 MA device (Tanita, Japan) | from enrollment to the end of the treatment/training at 14 weeks
  - skeletal muscle mass in kilograms
Anthropometric Measurements using TANITA MC-980 MA device (Tanita, Japan) | from enrollment to the end of treatment/training at 14 weeks
  * body fat mass in kilograms
  * body fat percentage (%)
Anthropometric Measurements using TANITA MC-980 MA device (Tanita, Japan) | from enrollment to the end of treatment/training at 14 weeks
  - fat free mass index based on weight, height and body fat percentage
Anthropometric Measurements using TANITA MC-980 MA device (Tanita, Japan) | from enrollment to the end of treatment/training at 14 weeks
  - visceral fat level 1-12: Healthy level of visceral fat. 13-59: Excessive level of visceral fat.
Anthropometric Measurements using Goniometer Saehen provide by StanleyMed | from enrollment to the end of treatment/training at 14 weeks
  Saehan Goniometr:
  - range of motion in the hip, knee and ankle joints (Adduction, Abduction, Flexion, Extension, External- and Internalrotation)
Anthropometric Measurement with SECA 201 anthropometric tape (SECA, Germany) | from enrollment to the end of treatment/training at 14 weeks
  - hip and waist circumferences
Anthropometric Measurements with SECA 201 anthropometric tape (SECA, Germany) | from enrollment to the end of treatment/training at 14 weeks
  - chest mobility
Anthropometric Measurement with SECA 201 anthropometric tape (SECA, Germany) | from enrollment to the end of treatment/training at 14 weeks
  - length and circumference of the lower limbs

CONTACTS AND LOCATIONS:
Overall Officials: Katarzyna Domaszewska, Prof.dr hab., Study Chair — University School of Physical Education in Poznan; Marta L Hofman, Master, Principal Investigator — The President Stanisław Wojciechowski State University of Applied Sciences in Kalisz; Piotr Szewczyk, Dr, Study Director — The President Stanisław Wojciechowski State University of Applied Sciences in Kalisz; Katarzyna Sobczak, Dr, Principal Investigator — University School of Physical Education in Poznan
Locations (1):
- The President Stanisław Wojciechowski State University of Applied Sciences in Kalisz, Kalisz, Wielkopolska, Poland

IPD SHARING:
Plan to Share IPD: Yes
in planning
Supporting Information: Study Protocol, SAP
Time Frame: Beginning 1 year after publication with no end date
Access Criteria: still on planning, beginning after the publication